CLINICAL TRIAL: NCT06187649
Title: A Systemic Review and Analysis of Factors and Outcomes in Breast Reconstruction
Brief Title: Infection After Implant-based Breast Reconstruction
Status: Active, not recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ung Sik Jin, Professor, Seoul National University Hospital
Other Study IDs: 2102-079-1197
Record Dates: First submitted 2023-12-18; First posted 2024-01-02 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Breast Implant Infection
MeSH Terms: interventions — Mammaplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: breast reconstruction — breast expander/implant insertion for breast reconstruction following mastectomy

SUMMARY:
Infections following postmastectomy breast reconstruction can compromise surgical outcomes and lead to significant morbidity. The aim of this study was to determine factors associated with infection following two-stage implant-based reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received implant-based breast reconstruction following mastectomy between 2015 and 2020 in Seoul National University Hospital

Exclusion Criteria:

* Patients who received flap surgery simultaneously with implant insertion

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Implant-based breast reconstruction following mastectomy
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Infection | 7 years
  Number of patients who developed requiring hospitalization-requiring infection

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ha JH, Ahn S, Kim HK, Lee HB, Moon HG, Han W, Hong KY, Chang H, Lee GK, Choi J, Jin US. Dynamic insights into infection risk over time in two-stage implant-based breast reconstruction: a retrospective cohort study. Int J Surg. 2024 Jun 1;110(6):3433-3439. doi: 10.1097/JS9.0000000000001235. PMID 38489664